CLINICAL TRIAL: NCT03619655
Title: Assessment of Multi-Modality Quantitative Imaging for Evaluation of Response of Metastatic Prostate Cancer to Therapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to changing prostate cancer standard of care, the research question became obsolete as the target population for the study no longer existed. The study is deemed not clinically relevant.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: J1835; IRB00165175 (Other: JHM IRB); U01CA140204 (NIH)
Record Dates: First submitted 2018-08-03; First posted 2018-08-08 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Prostate Cancer
Keywords: J1835; SPECT CT; PSMA; 18F-DCFPyL PET/CT; WB-MRI; NaF
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- "Cohort A" - SPECT CT and NaF PET (Experimental): Intervention 1: SPECT CT Intervention 2: NaF PET
  Interventions: Procedure: SPECT CT; Drug: 18F-NaF PET/CT
- "Cohort B" - SPECT CT and 18F-DCFPyL PET/CT (Experimental): Intervention 1: SPECT CT Intervention 2: 18F-DCFPyL PET/CT
  Interventions: Procedure: SPECT CT; Drug: 18F-DCFPyL PET/CT
- "Cohort C" - SPECT CT and WB-MRI (Experimental): Intervention 1: SPECT CT Intervention 2: WB-MRI
  Interventions: Procedure: SPECT CT; Procedure: WB-MRI

INTERVENTIONS:
Procedure: SPECT CT — MDP (99mTc-MDP) administration, about 180 min post-injection: whole body scan followed by a SPECT CT of regions designated by a board certified Nuclear Medicine physician after review of the whole body scan.
Drug: 18F-DCFPyL PET/CT — A bolus of ~9 mCi (333 MBq) of 18F-DCFPyL will be injected by slow IV push.
  Other Names: 18F-DCFPyL
  Arms: "Cohort B" - SPECT CT and 18F-DCFPyL PET/CT
Drug: 18F-NaF PET/CT — A dose of 5 mCi 18F-NaF is injected through the IV and followed by at least 10 ml of saline to flush the IV line of the remaining dose. At the 1 hour post injection time, total Whole Body Images take approximately 40 - 60 minutes depending on the height of the patient.
  Other Names: 18F-NaF; NaF PET
  Arms: "Cohort A" - SPECT CT and NaF PET
Procedure: WB-MRI — Whole body MRI exam (total examination time < 50 minutes)
  Other Names: Whole body MRI
  Arms: "Cohort C" - SPECT CT and WB-MRI

SUMMARY:
The study is an open label, non-randomized study designed to evaluate the diagnostic performance of SPECT CT.

DETAILED DESCRIPTION:
The study is an open label, non-randomized study designed to evaluate the diagnostic performance of SPECT CT. The study will consist of 3 cohorts, and a subset of the patients in cohort C will participate in a test-retest study, where the baseline SPECT/CT will be repeated.

SPECT CT will be performed in all cohorts.

Cohort A will evaluate SPECT CT by comparison to a Positron Emission Tomography (PET) scan using NaF.

Cohort B will evaluate SPECT CT by comparison to 18F-DCFPyL PET/CT.

Cohort C will evaluate SPECT CT by comparison to Whole Body Magnetic Resonance Imaging (WB-MRI).

Eligible subjects will be enrolled in a non-randomized manner per the treating physician discretion.

ELIGIBILITY:
Inclusion Criteria:

Males ≥18 years of age. Subjects provide signed informed consent and confirm that they are able and willing to comply with all protocol requirements.

Histologically confirmed adenocarcinoma of the prostate. Metastatic castration-resistant prostate cancer (mCRPC) with Bone metastases as manifested by one or more lesions on bone scan.

Documented castrate level of serum testosterone (≤50 ng/dl).

Documented progressive mCRPC based on at least one of the following criteria:

1. PSA progression defined as 25% increase over baseline value or nadir.
2. Radiographic progression for soft tissue lesions as per Response Evaluation Criteria in Solid Tumors (RECIST 1.1), and/ or radiographic progression for bone lesions as determined by radionuclide bone scan using the consensus guidelines of the PCWG3 criteria.

Planning to receive first line novel hormonal therapy with Abiraterone or Enzalutamide for the first time for mCRPC within 4 weeks of documented progression. Baseline scans will be obtained prior to starting new therapy.

Exclusion Criteria:

Subjects who are unable to give valid informed consent Subjects who are unwilling or unable to undergo an SPECT, PET or MR exam, including subjects with contra-indications to MR exams.

Subjects with prior Enzalutamide and Abiraterone for mCRPC Subjects with prior taxane chemotherapy for mCRPC Subjects administered any radioisotope within five physical half-lives or any IV X-ray contrast medium within 24 hours or any high density oral contrast medium (oral water contrast is acceptable) within 5 days prior to study drug injection.

Subjects with any medical condition or other circumstances that, in the opinion of the investigator, compromise obtaining reliable data, achieving study objectives, or completion.

Patients with a history reaction to gadolinium contrast agent. For cohort C, patients with renal failure (eGFR < 60ml/min/1.73m2) or patients on dialysis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Accuracy for Prediction of Progression Free Survival as determined by Quantitative bone SPECT indices (QBSIs) | Baseline, 3 months post-treatment, 6 months post-treatment, at time of disease progression assessed up to 5 years
  QBSI will be measured on SPECT scans at pre-defined intervals. A lower QBSI would mean likelier progression free survival.

SECONDARY OUTCOMES:
Reproducibility of the QBSIs using test-retest studies in 12 patients | 5 years
  Reproducibility measured by difference in QBSI between test-retest in 12 patients, as defined by the protocol. A smaller difference in QBSI reflects greater reproducibility.
Ability of QBSPECT to detect recurrence of metastatic disease as determined by QBSI in 60 patients. | Baseline, 3 months post-treatment, 6 months post-treatment, at time of disease progression assessed up to 5 years
  QBSI will be measured on QBSPECT images obtained at the same time as standard-of-care bone scans. A higher QBSI would predict earlier recurrence of metastasis.
Accuracy of NaF PET/CT as determined by difference in QBSI from SPECT versus QBSI from NaF PET/CT in 20 patients | Baseline, 3 months post-treatment, 6 months post-treatment, at time of disease progression assessed up to 5 years
  Difference in QBSI from SPECT versus NaF PET/CT. A smaller difference in the measured QBSI would reflect a higher accuracy of Na18F PET/CT. These images will be acquired within 32 hours of the bone scintigraphy scans at the pre-defined time points, per protocol.
Accuracy of PSMA PET/CT as determined by difference in QBSI from SPECT versus QBSI from PSMA PET/CT in 20 patients | Baseline, 6 months post-treatment, assessed up to 5 years
  Difference in QBSI from SPECT versus PSMA PET/CT. A smaller difference in the measured QBSI would reflect a higher accuracy of PSMA PET/CT. These images will be acquired within 32 hours of the bone scintigraphy scans at the pre-defined time points, per protocol.
Correlation of QBSI from SPECT/CT to restricted diffusion obtained from whole body MRI | 5 years
  Ratio of QBSI obtained from SPECT imaging to quantitative biomarkers of restricted diffusion (diffusion-weighted imaging) obtained from a WB-MRI protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Lilja Solnes, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No